CLINICAL TRIAL: NCT00710710
Title: An Open, Randomised, Clinical Phase II Trial in Patients With Unresectable Advanced Pancreatic Cancer Investigating the Efficacy, Safety, and Pharmacokinetics of BI 2536 Administered in Repeated 3-week Cycles as a Single i.v. Dose of 200 mg on Day 1 or as 60 mg Doses on Days 1, 2, and 3
Brief Title: Open, Randomized Phase II Trial to Investigate the Efficacy and Safety of the PLK-1 Inhibitor BI 2536 in Patients With Advanced, Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1216.10
Record Dates: First submitted 2008-07-03; First posted 2008-07-04 (Estimated); Results first posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — BI 2536

ARMS (2):
- BI 2536 High dose (Experimental): Day 1
  Interventions: Drug: BI 2536
- BI 2536 Low dose (Experimental): Day 1 - 3
  Interventions: Drug: BI 2536

INTERVENTIONS:
Drug: BI 2536 — Intravenous Infusion

SUMMARY:
The trial is conducted in order to evaluate the efficacy, safety and pharmacokinetics of BI 2536 in the treatment of unresectable advanced pancreatic cancer as first line or second line therapy. A secondary aim is to identify the most suitable dosage regimen for the further phase II and III clinical programme of BI 2536. To achieve this objective, two dosage regimens are compared in patients receiving first line therapy.

ELIGIBILITY:
Inclusion Criteria:

1. male or female patient aged 18 years or older
2. patient with confirmed diagnosis of unresectable, either locally advanced or metastatic, ductal adenocarcinoma of the pancreas
3. patient who is either chemonaïve (for the first line cohorts), or who presents with progressive disease under first line chemotherapy with a gemcitabine based regimen (for the second line cohort)
4. Karnofsky performance status of ¿ 70% for the first line cohorts, and Karnofsky performance status ¿ 50% for the second line cohort
5. patient with at least one measurable tumour lesion that can accurately be measured by magnetic resonance imaging (MRI), or computed tomography (CT) in at least one dimension (longest diameter to be recorded)
6. life expectancy of at least three months
7. patient must have given written informed consent consistent with the guidelines of the international conference on harmonisation for good clinical practice (ICH-GCP) as well as with local legislation

Exclusion Criteria:

1. prior adjuvant chemotherapy (for first line cohorts only)
2. ampullary carcinoma of the pancreas
3. hypersensitivity to the trial drug or the excipients
4. persistence of toxicities of prior anti cancer therapies which are deemed to be clinically relevant
5. known second malignancy requiring therapy
6. brain metastases which are symptomatic or require therapy
7. absolute neutrophil count less than 1.500/mm3
8. platelet count less than 100.000/mm3
9. haemoglobin less than 9 mg/dl
10. aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 2.5 times the upper limit of normal, or AST or ALT greater than 5 times the upper limit of normal in case of known liver metastases
11. bilirubin greater than 3.0 mg/dl (> 52 ¿mol/l, SI unit equivalent) under adequate drainaging measures (in case of obstructive jaundice)
12. serum creatinine greater than 2.0 mg/dl
13. concomitant intercurrent illnesses including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness or social situation that would limit compliance with trial requirement or which are considered relevant for the evaluation of the efficacy or safety of the trial drug
14. radiotherapy within the past four weeks prior to treatment with the trial drug
15. hormone- or immunotherapy or therapy with a biologic response modifier within the past four weeks
16. treatment with any other investigational drug within the past four weeks
17. men or women who are sexually active and unwilling to use a medically acceptable method of contraception (e.g. abstinence, condom with spermicidal coating, diaphragm with spermicidal coating, oral contraceptive, progesterone implant, sterilisation) during the trial
18. pregnancy or lactation
19. patients unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2006-08-01 (Actual); Primary Completion 2008-10-14 (Actual); Study Completion 2008-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (10):
- 1216.10.43001 Boehringer Ingelheim Investigational Site, Vienna, Austria
- Germany (9):
  - 1216.10.49013 Boehringer Ingelheim Investigational Site, Celle
  - 1216.10.49009 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1216.10.49007 Boehringer Ingelheim Investigational Site, Essen
  - 1216.10.49001 Boehringer Ingelheim Investigational Site, Freiburg/Breisgau
  - 1216.10.49005 Boehringer Ingelheim Investigational Site, Hamburg
  - 1216.10.49010 Boehringer Ingelheim Investigational Site, Herne
  - 1216.10.49008 Boehringer Ingelheim Investigational Site, München
  - 1216.10.49003 Boehringer Ingelheim Investigational Site, Stuttgart
  - 1216.10.49002 Boehringer Ingelheim Investigational Site, Ulm

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was an open, randomised, clinical phase II trial in patients with unresectable advanced pancreatic cancer investigating the efficacy, safety, and pharmacokinetics of BI 2536 administered in repeated 3-week cycles as a single IV dose of 200 mg on Day 1 or as 60 mg doses on Days 1, 2, and 3
Pre-assignment Details: Only subjects that met all the study inclusion and none of the exclusion criteria were to be entered in the study.
Groups:
- 200mg BI 2536 IV on Day 1: 200 milligram (mg) given as an intravenous (IV) infusion on day 1 of each 3 week cycle, to a total dose of 200 mg. Each patient was to receive at least 2 treatment courses. In the case of benefit (i.e. at least stable disease and acceptable tolerability), the patient could continue therapy with the trial drug.
- 60mg BI 2536 IV on Day 1-3: 60 milligram (mg) given as an intravenous (IV) infusion on day 1, 2 and 3 of each 3 week cycle. Each patient was to receive at least 2 treatment courses. In the case of benefit (i.e. at least stable disease and acceptable tolerability), the patient could continue therapy with the trial drug.
Period: Overall Study
Arm/Group | 200mg BI 2536 IV on Day 1 | 60mg BI 2536 IV on Day 1-3
Started | 45 | 44
Treated | 43 | 43
Completed | 0 | 0
Not Completed | 45 | 44
Not completed — Consent withdrawn | 2 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 3 | 3
Not completed — Progressive disease | 40 | 38

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): all patients who received at least 1 single dose of BI 2536 were considered, including patients who had been replaced for any reason.
Groups:
- Total: Total of all reporting groups
Arm/Group | 200mg BI 2536 IV on Day 1 | 60mg BI 2536 IV on Day 1-3 | Total
Number analyzed (Participants) | 43 | 43 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (9.4) | 63.0 (9.3) | 63.3 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 30 | 29 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 43 | 43 | 86
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Quality of Life: Overall health [Mean (Standard Deviation); unit: Score on a scale] — Quality of life (QOL) was measured using the widely used and validated measure the European Organization for Research and Treatment - Quality of Life Questionnaire (EORTC QLQ-C30), based on questions 29 "How would you rate your overall health during the past week?" and 30 "How would you rate your overall quality of life during the past week?", scored between 1 (very poor) to 7 (Excellent).
  Score on a scale | 3.8 (1.21) | 4.1 (1.31) | 4.0 (1.26)
Quality of Life: Quality of life [Mean (Standard Deviation); unit: Score on a scale] — Quality of life (QOL) was measured using the widely used and validated measure the European Organization for Research and Treatment - Quality of Life Questionnaire (EORTC QLQ-C30), based on questions 29 "How would you rate your overall health during the past week?" and 30 "How would you rate your overall quality of life during the past week?", scored between 1 (very poor) to 7 (Excellent).
  Score on a scale | 3.8 (1.51) | 4.3 (1.40) | 4.0 (1.47)

OUTCOME MEASURES:

1. Primary Outcome: Best Objective Response Evaluated According to the RECIST Criteria by Independent Review
Description: Best objective response: Tumour assessment by independent review of tumour imaging by an external contract research organization (CRO) according to Response Evaluation Criteria In Solid Tumours (RECIST) after every second treatment course, including imaging (e.g. Computed tomography (CT), Magnetic resonance imaging (MRI)) and submission of image(s) to central imaging unit.
  Complete remission (CR): Disappearance of all target lesions for at least 4 weeks from the documentation of CR.
  Partial remission (PR): At least a 30% decrease in the sum of LD of target lesions taking as reference the baseline sum Longest Diameter (LD).
  Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as references the smallest sum LD since the treatment started.
  No best response: includes all RECIST categories which are considered as failing to respond to therapy, e.g. progressive disease, death or unknown.
Time Frame: Tumour measurements performed at screening (day -21 to -1), at the end of every other treatment period (2x 3 weeks), and at the end of the trial or when a patient concluded the trial, up to 357 days.
Population: Treated Set (TS): all patients who received at least 1 single dose of BI 2536 and who had an evaluation after baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | 200mg BI 2536 IV on Day 1 | 60mg BI 2536 IV on Day 1-3
Number analyzed (Participants) | 34 | 36
Participants
  Confirmed best overall response: Complete response | 0 | 0
  Confirmed best overall response: Partial response | 1 | 1
  Confirmed best overall response: Stable disease | 11 | 10
  Confirmed best overall response: No best response | 22 | 25
  Unconfirmed best overall response: Complete response | 0 | 0
  Unconfirmed best overall response: Partial response | 1 | 2
  Unconfirmed best overall response: Stable disease | 20 | 18
  Unconfirmed best overall response: No best response | 13 | 16
Statistical Analysis 1: Comparison: 200mg BI 2536 IV on Day 1; Confirmed objective response, comparison with historical controls (Gemcitabine); Test type: Other; p = 0.7021, Exact binomial test — p0 = 0.056, one sided exact binomial test with a 2.5% significance level; Maximum likelihood estimation = 0.0233, 95% CI 2-sided [0.0006 to 0.1229]
Statistical Analysis 2: Comparison: 200mg BI 2536 IV on Day 1; Confirmed objective response, comparison with historical controls (Gemcitabine); Test type: Other; p = 0.9156, Exact binomial test — p0 = 0.092, one sided exact binomial test with a 2.5% significance level; Maximum likelihood estimation = 0.0233, 95% CI 2-sided [0.0006 to 0.1229]
Statistical Analysis 3: Comparison: 60mg BI 2536 IV on Day 1-3; Confirmed objective response, comparison with historical controls (Gemcitabine); Test type: Other; p = 0.7021, Exact binomial test — p0 = 0.056, one sided exact binomial test with a 2.5% significance level; Maximum likelihood estimation = 0.0233, 95% CI 2-sided [0.0006 to 0.1229]
Statistical Analysis 4: Comparison: 60mg BI 2536 IV on Day 1-3; Confirmed objective response, comparison with historical controls (Gemcitabine); Test type: Other; p = 0.9156, Exact binomial test — p0 = 0.092, one sided exact binomial test with a 2.5% significance level; Maximum likelihood estimation = 0.0233, 95% CI 2-sided [0.0006 to 0.1229]

2. Secondary Outcome: Tumour Control After the Fourth Treatment Course
Description: Tumour control rate was defined as the number of patients in a treatment arm who had completed 4 courses of treatment and presented with Stable Disease (SD), Partial Response (PR), or Complete Remission (CR). Tumour assessment by independent review of tumour imaging according to RECIST after every second treatment course, including imaging (e.g. CT, MRI) and submission of image(s) to central imaging unit.
  Complete remission (CR): Disappearance of all target lesions for at least 4 weeks from the documentation of CR.
  Partial remission (PR): At least a 30% decrease in the sum of LD of target lesions taking as reference the baseline sum Longest Diameter (LD).
  Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as references the smallest sum LD since the treatment started.
  The secondary endpoint "duration of overall response" was integrated into and displayed with tumour control endpoints.
Time Frame: Tumour measurements performed at screening (day -21 to -1) and at the end of of the fourth 3-week treatment cycle, up to 105 days.
Population: Treated Set (TS): all patients who received at least 1 single dose of BI 2536 and who had an evaluation after baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | 200mg BI 2536 IV on Day 1 | 60mg BI 2536 IV on Day 1-3
Number analyzed (Participants) | 43 | 43
Participants
  Tumour control: yes | 7 | 4
  Tumour control: no | 14 | 19
  Tumour control: unknown | 22 | 20

3. Secondary Outcome: Duration of Overall Response
Description: The duration of overall response was measured from the time measurement criteria were met for complete remission (CR) or partial remission (PR) (whichever was first recorded) until the first date that recurrent or progressive disease was objectively documented, taking as reference for progressive disease the smallest measurements recorded since the treatment started.
  Tumour assessment by independent review of tumour imaging by an external CRO according to RECIST after every second treatment course, including imaging (e.g. CT, MRI) and submission of image(s) to central imaging unit.
Time Frame: as for outcome 1
Population: All patients who received at least 1 single dose of BI 2536, who had an evaluation after baseline and who had an unconfirmed best overall response by independent review.
Measure: Median (Standard Deviation); unit: Days
Arm/Group | 200mg BI 2536 IV on Day 1 | 60mg BI 2536 IV on Day 1-3
Number analyzed (Participants) | 1 | 2
Days | 42 (NA) — Data available for only one subject, dispersion value not calculable. | 141 (138.59)

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) was defined as the duration of time from randomisation to time of progression or death. For patients without documented progression at the time of analysis, PFS was censored as the total observation time without new anti-cancer therapy. PFS was analysed with the Kaplan-Meier method for each of the treatment arms. Kaplan-Meier estimates and confidence intervals were tabulated at specific points in time. Greenwood's variance estimate was used to form confidence intervals.
  Progressive disease: At least a 20% increase in the sum of Longest Diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 200mg BI 2536 IV on Day 1 | 60mg BI 2536 IV on Day 1-3
Number analyzed (Participants) | 43 | 43
days | 47 [43 to 87] | 46 [43 to 56]
Statistical Analysis 1: Comparison: 200mg BI 2536 IV on Day 1 vs 60mg BI 2536 IV on Day 1-3; Test type: Other; p = 0.38, Regression, Cox; Hazard Ratio (HR) = 1.22, 95% CI 2-sided [0.78 to 1.91] — if HR is below 1, then 60mg BI 2536 IV on day 1-3 is better

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was the time from first treatment until death. If there was no occurrence of death or progression until the last follow-up of the trial, the time was to be censored at the date of last trial visit. OS was analysed with the Kaplan-Meier method for each of the treatment arms. Kaplan-Meier estimates and confidence intervals were tabulated at specific points in time. Greenwood's variance estimate was used to form confidence intervals.
  The secondary endpoint "One-year survival" was integrated into the secondary endpoint overall survival.
Time Frame: From first treatment till the end of the trial or when a patient concluded the trial, up to 336 days.
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 200mg BI 2536 IV on Day 1 | 60mg BI 2536 IV on Day 1-3
Number analyzed (Participants) | 43 | 43
days | 154 [103 to 302] | 148 [81 to 315]
Statistical Analysis 1: Comparison: 200mg BI 2536 IV on Day 1 vs 60mg BI 2536 IV on Day 1-3; Test type: Other; p = 0.69, Regression, Cox; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.68 to 1.78] — if HR is below 1, then 60mg BI 2536 IV on day 1-3 is better

6. Secondary Outcome: Best Objective Response Evaluated According to the RECIST Criteria by Investigator Assessment
Description: Best objective response: Tumour assessment by investigator assessment of tumour imaging according to Response Evaluation Criteria In Solid Tumours (RECIST) after every second treatment course, including imaging (e.g. Computed tomography (CT), Magnetic resonance imaging (MRI)) and submission of image(s) to central imaging unit.
  Complete remission (CR): Disappearance of all target lesions for at least 4 weeks from the documentation of CR.
  Partial remission (PR): At least a 30% decrease in the sum of LD of target lesions taking as reference the baseline sum Longest Diameter (LD).
  Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as references the smallest sum LD since the treatment started.
  No best response: includes all RECIST categories which are considered as failing to respond to therapy, e.g. progressive disease, death or unknown.
Time Frame: as for outcome 1
Population: Treated Set (TS): all patients who received at least 1 single dose of BI 2536 were considered, including patients who had been replaced for any reason. 4 patients did not have any evaluations after baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | 200mg BI 2536 IV on Day 1 | 60mg BI 2536 IV on Day 1-3
Number analyzed (Participants) | 39 | 43
Participants
  Confirmed best overall response: Complete response | 0 | 0
  Confirmed best overall response: Partial response | 0 | 0
  Confirmed best overall response: Stable disease | 11 | 11
  Confirmed best overall response: No best response | 28 | 32
  Unconfirmed best overall response: Complete response | 0 | 0
  Unconfirmed best overall response: Partial response | 0 | 0
  Unconfirmed best overall response: Stable disease | 36 | 38
  Unconfirmed best overall response: No best response | 3 | 5
Statistical Analysis 1: Comparison: 200mg BI 2536 IV on Day 1; Confirmed objective response, comparison with historical controls (Gemcitabine); Test type: Other; p = 0.9161, Exact binomial test — p0 = 0.056, one sided exact binomial test with a 2.5% significance level; Maximum likelihood estimation = 0, 95% CI 2-sided [0.0000 to 0.0822]
Statistical Analysis 2: Comparison: 200mg BI 2536 IV on Day 1; Confirmed objective response, comparison with historical controls (Gemcitabine); Test type: Other; p = 0.9842, Exact binomial test — p0 = 0.092, one sided exact binomial test with a 2.5% significance level; Maximum likelihood estimation = 0, 95% CI 2-sided [0.0000 to 0.0822]
Statistical Analysis 3: Comparison: 60mg BI 2536 IV on Day 1-3; Confirmed objective response, comparison with historical controls (Gemcitabine); Test type: Other; p = 0.9161, Exact binomial test — p0 = 0.056, one sided exact binomial test with a 2.5% significance level; Maximum likelihood estimation = 0, 95% CI 2-sided [0.0000 to 0.0822]
Statistical Analysis 4: Comparison: 60mg BI 2536 IV on Day 1-3; Confirmed objective response, comparison with historical controls (Gemcitabine); Test type: Other; p = 0.9842, Exact binomial test — p0 = 0.092, one sided exact binomial test with a 2.5% significance level; Maximum likelihood estimation = 0, 95% CI 2-sided [0.0000 to 0.0822]

7. Secondary Outcome: One-year Survival
Description: One-year survival was defined as survival at 1 year after randomisation. For the cohort of first line patients, this time point coincided with the beginning of treatment with the Trial drug. For second line patients, 1 year survival was defined as 1 year after the start of the previous first line treatment for pancreatic cancer.
Time Frame: 1 year, see description for detailed definition of the time frame.
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | 200mg BI 2536 IV on Day 1 | 60mg BI 2536 IV on Day 1-3
Number analyzed (Participants) | 43 | 43
participants | 4 | 5

8. Secondary Outcome: Number of Participants With Carbohydrate Antigen 19-9 (CA19-9) Response
Description: Number of participants with carbohydrate antigen 19-9 (CA19-9) response rate was defined as the proportion of patients with a decrease in CA19-9 serum levels of ≥25% from baseline in 2 consecutive measurements performed ≥4 weeks apart. Additionally, the proportion of patients with an improved response was assessed, i.e. a decrease in CA19-9 of ≥75% at 2 consecutive measurements ≥4 weeks apart. By definition, a positive CA19-9 response could not occur in patients with normal baseline CA19-9 levels.
Time Frame: Blood samples for CA19-9 analysis were collected on Days 1, 2, and 5 of each treatment period, up to 357 days.
Population: Treated Set (TS): all patients who received at least 1 single dose of BI 2536 were considered, including patients who had been replaced for any reason. 19 patients did not have elevated CA19-9 levels at baseline and could not be included.
Measure: Count of Participants; unit: Participants
Arm/Group | 200mg BI 2536 IV on Day 1 | 60mg BI 2536 IV on Day 1-3
Number analyzed (Participants) | 43 | 43
Participants
  CA19-9 response: No | 41 | 41
  CA19-9 response: Yes | 2 | 2
  Improved CA19-9 response: No | 43 | 43
  Improved CA19-9 response: Yes | 0 | 0

9. Secondary Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Description: Dose limiting toxicity (DLT) was defined as drug-related CTCAE (Common Terminology Criteria for Adverse Events, version 3.0) grade ≥3 non-haematological toxicity (excluding untreated nausea, vomiting or diarrhoea), drug related CTCAE grade 4 neutropenia for ≥7 days and / or complicated by infection of CTCAE grade 4, or drug related CTCAE grade 4 haematological toxicity other than neutropenia.
Time Frame: as for outcome 1
Population: Treated Set (TS): all patients who received at least 1 single dose of BI 2536 were considered, including patients who had been replaced for any reason. 1 participants did not experience any adverse event and was not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 200mg BI 2536 IV on Day 1 | 60mg BI 2536 IV on Day 1-3
Number analyzed (Participants) | 43 | 42
Participants
  No | 32 | 27
  Yes | 11 | 15

10. Secondary Outcome: Quality of Life Assessment, Including Clinical Benefit Response: Overall Health
Description: Quality of life (QOL) was measured using the widely used and validated measure the European Organization for Research and Treatment - Quality of Life Questionnaire (EORTC QLQ-C30), based on questions 29 "How would you rate your overall health during the past week?" and 30 "How would you rate your overall quality of life during the past week?", scored between 1 (very poor) to 7 (Excellent).
Time Frame: Data from the last available questionnaire for each patient. Questionnaires were taken at screening (day -21 to -1), at the beginning (Day 1) and end (Day 22 ± 3) of every treatment period (3 weeks), and at the end of the trial, up to 357 days.
Population: Treated Set (TS): all patients who received at least 1 single dose of BI 2536 and who had an evaluation after baseline.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 200mg BI 2536 IV on Day 1 | 60mg BI 2536 IV on Day 1-3
Number analyzed (Participants) | 39 | 40
Score on a scale | 3.8 (1.17) | 4.1 (1.41)

11. Secondary Outcome: Quality of Life Assessment, Including Clinical Benefit Response: Quality of Life
Description: as for outcome 10
Time Frame: as for outcome 10
Population: Treated Set (TS): all patients who received at least 1 single dose of BI 2536 and who had an evaluation after baseline.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 200mg BI 2536 IV on Day 1 | 60mg BI 2536 IV on Day 1-3
Number analyzed (Participants) | 38 | 40
Score on a scale | 3.8 (1.29) | 4.2 (1.45)

12. Secondary Outcome: Number of Participants With Incidence and Intensity of Adverse Events Graded According to Common Terminology Criteria for Adverse Events (CTCAE)
Description: Number of participants with incidence and intensity of Adverse Events (AE) graded according to CTCAE. Intensity of AEs was scaled according to US-NCI CTCAE, version 3.0. Severity grades 1 to 5 were based on the following general guidelines, with unique clinical descriptions of severity for each AE:
  * Grade 1 Mild
  * Grade 2 Moderate
  * Grade 3 Severe
  * Grade 4 Life-threatening or disabling
  * Grade 5 Death
Time Frame: From first administration until 21 days after the day of last administration, up to 16 cycles, up to 357 days.
Population: Treated Set (TS): all patients who received at least 1 single dose of BI 2536 were considered, including patients who had been replaced for any reason. 1 patient did not experience any AE and was not included in the endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | 200mg BI 2536 IV on Day 1 | 60mg BI 2536 IV on Day 1-3
Number analyzed (Participants) | 43 | 42
Participants
  Grade 1 | 5 | 5
  Grade 2 | 7 | 4
  Grade 3 | 12 | 16
  Grade 4 | 9 | 9
  Grade 5 | 10 | 8

ADVERSE EVENTS:
Time Frame: from first administration until 21 days after the day of last administration, up to 16 cycles, up to 357 days.
Description: Treated Set (TS): all patients who received at least 1 single dose of BI 2536 were considered, including patients who had been replaced for any reason.
Arm/Group | 200mg BI 2536 IV on Day 1 | 60mg BI 2536 IV on Day 1-3
All-Cause Mortality (participants affected / at risk) | 32/43 | 35/43
Serious Adverse Events (participants affected / at risk) | 22/43 | 23/43
Other Adverse Events (participants affected / at risk) | 41/43 | 41/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 200mg BI 2536 IV on Day 1 (N=43) | 60mg BI 2536 IV on Day 1-3 (N=43)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Anal fissure (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 2 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2
Subileus (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 1 | 2
General physical health deterioration (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 2
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 2 | 1
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Biliary sepsis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 3 | 2
Pneumonia (Infections and infestations) | 4 | 4
Sepsis (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Device dislocation (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 5
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral artery embolism (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bile duct stent insertion (Surgical and medical procedures) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 200mg BI 2536 IV on Day 1 (N=43) | 60mg BI 2536 IV on Day 1-3 (N=43)
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Leukopenia (Blood and lymphatic system disorders) | 14 | 9
Neutropenia (Blood and lymphatic system disorders) | 17 | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 4
Abdominal pain (Gastrointestinal disorders) | 8 | 6
Abdominal pain upper (Gastrointestinal disorders) | 3 | 5
Ascites (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 13 | 10
Diarrhoea (Gastrointestinal disorders) | 10 | 9
Dry mouth (Gastrointestinal disorders) | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 6 | 5
Dysphagia (Gastrointestinal disorders) | 0 | 3
Flatulence (Gastrointestinal disorders) | 10 | 7
Nausea (Gastrointestinal disorders) | 13 | 18
Vomiting (Gastrointestinal disorders) | 14 | 8
Asthenia (General disorders) | 1 | 3
Fatigue (General disorders) | 17 | 23
Oedema peripheral (General disorders) | 4 | 5
Pain (General disorders) | 1 | 5
Pyrexia (General disorders) | 3 | 7
Urinary tract infection (Infections and infestations) | 2 | 3
Drug administration error (Injury, poisoning and procedural complications) | 1 | 3
Blood alkaline phosphatase increased (Investigations) | 3 | 0
Haemoglobin decreased (Investigations) | 5 | 8
Weight decreased (Investigations) | 1 | 5
Anorexia (Metabolism and nutrition disorders) | 8 | 14
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 8
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Dizziness (Nervous system disorders) | 8 | 5
Polyneuropathy (Nervous system disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 3 | 4
Sleep disorder (Psychiatric disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Hypertension (Vascular disorders) | 2 | 4
Hypotension (Vascular disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.